CLINICAL TRIAL: NCT04767438
Title: STUDY PROTOCOL FOR A PROSPECTIVE, MULTICENTRE, COHORT STUDY: Preeclampsia Sequential Screening Using Angiogenic Factors During First Trimester of Pregnancy (CRISP STUDY)
Brief Title: Preeclampsia Sequential Screening Using Angiogenic Factors During First Trimester of Pregnancy
Acronym: CRISP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Daniel Orós López, Fetal Medicine, Associate Professor, University of Zaragoza, Instituto de Investigación Sanitaria Aragón
Other Study IDs: CRISP
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Pre-Eclampsia; Pregnancy Complications
Keywords: Preeclampsia; Screening
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: All singleton pregnancies that present to the 12-week scan in the Obstetrics Unit of the participant hospitals. Singleton pregnancies; Gestational age less than 14 weeks, estimated according to Crown-Rump Length (CRL); Blood sample between 8 and 14 weeks of pregnancy; Patients who accept to participate in the study and sign the informed consent.
  Interventions: Other: Pregnant women

INTERVENTIONS:
Other: Pregnant women — All pregnant women that present to the 12-week scan in the Obstetrics Unit

SUMMARY:
Preeclampsia (PE) affects from 2 to 8% of pregnant women. Recent studies show that prevention is the best strategy to improve perinatal outcomes. Therefore, the development of new strategies for preeclampsia screening becomes essential in order to determine the individual risk for each patient, and thus, to identify those who would be candidates for receiving prophylactic treatment with low-dose aspirin from the first trimester of pregnancy. The aim of our study is to determine prospectively, during clinical practice, the predictive and preventive capacity of a model of preeclampsia sequential screening in the first trimester of pregnancy.

This is a prospective, multicentre, cohort study, with the collaboration of Hospital de la Santa Creu i Sant Pau (Barcelona), Hospital Universitario de Cruces (Bilbao), Hospital Son Llàtzer (Mallorca) and Hospital Clínico Universitario Lozano Blesa (Zaragoza). Women with a singleton pregnancy attending to the 12-week ultrasound scan at one of the maternity hospitals participating in the study between March 1st 2021 and 30th October 2021 will be recruited. Patients who accept to participate in the study will be classified into three risk groups (low-risk, moderate-risk and high risk) based on medical history, Mean Arterial Pressure (MAP), Pregnancy-Associated Plasma Protein A (PAPP-A) and Uterine Artery Pulsatility Index (UTPI). Placental Growth Factor (PlGF) will only be determined in those patients classified as intermediate risk after this first step and then reclassified in high and low-risk patients depending on its values. The number of first-trimester scans performed by these hospitals is approximately 8200 patients annually. Due to PE prevalence in our environment is around 3% of the total population, a total of 246 cases of PE are to be expected. Therefore, based on similar previous experiences, we could assume that 80% of the patients will accept to participate in the study, meaning a total sample of 6560 pregnant women.

DETAILED DESCRIPTION:
All the data required to carry out this study, including those derived from sonographies and blood tests, will be collected during the normal pregnancy control, without further appointments. A blood test will be requested in all pregnant women in the first appointment of pregnancy control between 9 and 13 weeks, to determine risk of chromosomal disorders according to the national protocol and it will be used this same sample to analyze angiogenic factors without requiring new blood extractions. In the first-trimester scan, the mean uterine arteries pulsatility index will be determined, as well as mean arterial pressure. In this visit, the patient will be asked about her medical history. We will offer the patients the inclusion to our study in that moment; those who agree to participate in the study will sign the informed consent. In the participants, the initial risk of PE will be calculated using maternal medical history, MAP, UTPI and PAPP-A (already used in aneuploidies screening), using the software validated to each laboratory. Patients will be classified into 3 groups:

* Low risk of PE (<1/500)
* Intermediate risk of PE (between 1/50 and 1/500)
* High risk of PE (>1/50) In those patients classified as intermediate and high-risk, PlGF and s-Flt-1 will be determined from the blood samples kept in biobanks of each hospital according to the current legislation. SFlt-1 results will be analyzed at the end of the study in order to decrease the cost because there will not be used to make clinical decisions. PlGF in high-risk patients will not be considered either to reclassify those patients. In both cases, the diagnostic efficiency will be analyzed at the end of the study.

Patients in the intermediate-risk group (1/50-1/500) will be reclassified after adding PlGF levels in the predictive algorithm in 2 groups: Low risk of PE (<1/160) and High risk of PE (>1/160).

To the patients classified as high risk at any of the steps, will be offered prophylactic treatment with AcetylSalicylic acid (ASA) (150mg/24h) until 36 weeks of pregnancy, if there is not a contraindication. All data from eligible patients will be analyzed. A bivariant statistical analysis will be performed in order to assess the relationship between dependent variables (diagnose of PE and/or IUGR) and the other variables included in this study

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies;
* Gestational age less than 14 weeks, estimated according to Crown-Rump Length (CRL);
* Blood sample between 8 and 14 weeks of pregnancy;
* Patients who accept to participate in the study and sign the informed consent

Exclusion Criteria:

* Fetus with chromosomal disorders, major congenital malformations or congenital infections diagnosed in the first-trimester ultrasound;
* Multiple pregnancies;
* Non-acceptance of participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every singleton pregnancy attending during the period study
Sampling Method: Non-Probability Sample
Enrollment: 6560 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of preeclampsia | 30 weeks
  Diagnosis of preeclampsia during pregnancy following the definition of the International Society for the Study of Hypertension in Pregnancy, (ISSHP)

SECONDARY OUTCOMES:
Early-onset Preeclampsia | 30 weeks
  Early-onset Preeclampsia: diagnosos before 34 weeks of pregnancy
Severe preeclampsia | 30 weeks
  Severe preeclampsia (ISSHP)
Pregnancy-induced hypertension | 30 weeks
  Pregnancy-induced hypertension
SGA | 30 weeks
  Small for gestational age: birth weight below the 10th percentile
IUGR | 30 weeks
  Intrauterine Growth Restriction
Perinatal mortality | 30 weeks
  Perinatal mortality (>22 weeks of pregnancy - < 28 days postpartum)
Neonatal acidosis | 30 weeks
  Neonatal acidosis (arterial pH <7.10 + base excess >12mEq/L)
Neonatal Intensive Care Unit | 16 weeks
  Days of admission in neonatal Intensive Care Unit
Neonatal morbidity | 16 weeks
  Significant neonatal morbidity: convulsions, intraventricular haemorrhage > III grade, periventricular leukomalacia, hypoxic-ischemic encephalopathy, abnormal electroencephalogram, necrotizing enterocolitis, acute renal failure (serum creatinine >1.5mg/dL) or heart failure (requiring inotropic agents).
Gestational age at birth | 30 weeks
  Gestational age at birth
Type of delivery | 30 weeks
  Type of delivery (vaginal, spontaneous or instrumental, cesarean section)
Cost of the analysis of angiogenic and antiangiogenic factors | 18 months
  The economic cost of the analysis of angiogenic and antiangiogenic factors in euros (PlGF and sFlt-1).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duley L. The global impact of pre-eclampsia and eclampsia. Semin Perinatol. 2009 Jun;33(3):130-7. doi: 10.1053/j.semperi.2009.02.010. PMID 19464502
- [Background] Melchiorre K, Wormald B, Leslie K, Bhide A, Thilaganathan B. First-trimester uterine artery Doppler indices in term and preterm pre-eclampsia. Ultrasound Obstet Gynecol. 2008 Aug;32(2):133-7. doi: 10.1002/uog.5400. PMID 18615872
- [Background] Lisonkova S, Sabr Y, Mayer C, Young C, Skoll A, Joseph KS. Maternal morbidity associated with early-onset and late-onset preeclampsia. Obstet Gynecol. 2014 Oct;124(4):771-781. doi: 10.1097/AOG.0000000000000472. PMID 25198279
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] von Beckerath AK, Kollmann M, Rotky-Fast C, Karpf E, Lang U, Klaritsch P. Perinatal complications and long-term neurodevelopmental outcome of infants with intrauterine growth restriction. Am J Obstet Gynecol. 2013 Feb;208(2):130.e1-6. doi: 10.1016/j.ajog.2012.11.014. Epub 2012 Nov 15. PMID 23159694
- [Background] Melamed N, Klinger G, Tenenbaum-Gavish K, Herscovici T, Linder N, Hod M, Yogev Y. Short-term neonatal outcome in low-risk, spontaneous, singleton, late preterm deliveries. Obstet Gynecol. 2009 Aug;114(2 Pt 1):253-260. doi: 10.1097/AOG.0b013e3181af6931. PMID 19622985
- [Background] Escobar GJ, Clark RH, Greene JD. Short-term outcomes of infants born at 35 and 36 weeks gestation: we need to ask more questions. Semin Perinatol. 2006 Feb;30(1):28-33. doi: 10.1053/j.semperi.2006.01.005. PMID 16549211
- [Background] Phipps EA, Thadhani R, Benzing T, Karumanchi SA. Pre-eclampsia: pathogenesis, novel diagnostics and therapies. Nat Rev Nephrol. 2019 May;15(5):275-289. doi: 10.1038/s41581-019-0119-6. PMID 30792480
- [Background] Flint EJ, Cerdeira AS, Redman CW, Vatish M. The role of angiogenic factors in the management of preeclampsia. Acta Obstet Gynecol Scand. 2019 Jun;98(6):700-707. doi: 10.1111/aogs.13540. Epub 2019 Feb 22. PMID 30667052
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Roberge S, Bujold E, Nicolaides KH. Aspirin for the prevention of preterm and term preeclampsia: systematic review and metaanalysis. Am J Obstet Gynecol. 2018 Mar;218(3):287-293.e1. doi: 10.1016/j.ajog.2017.11.561. Epub 2017 Nov 11. PMID 29138036
- [Background] Wright D, Rolnik DL, Syngelaki A, de Paco Matallana C, Machuca M, de Alvarado M, Mastrodima S, Tan MY, Shearing S, Persico N, Jani JC, Plasencia W, Papaioannou G, Molina FS, Poon LC, Nicolaides KH. Aspirin for Evidence-Based Preeclampsia Prevention trial: effect of aspirin on length of stay in the neonatal intensive care unit. Am J Obstet Gynecol. 2018 Jun;218(6):612.e1-612.e6. doi: 10.1016/j.ajog.2018.02.014. Epub 2018 Mar 2. PMID 29505771
- [Background] Roberge S, Villa P, Nicolaides K, Giguere Y, Vainio M, Bakthi A, Ebrashy A, Bujold E. Early administration of low-dose aspirin for the prevention of preterm and term preeclampsia: a systematic review and meta-analysis. Fetal Diagn Ther. 2012;31(3):141-6. doi: 10.1159/000336662. Epub 2012 Mar 21. PMID 22441437
- [Background] Bujold E, Roberge S, Lacasse Y, Bureau M, Audibert F, Marcoux S, Forest JC, Giguere Y. Prevention of preeclampsia and intrauterine growth restriction with aspirin started in early pregnancy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):402-414. doi: 10.1097/AOG.0b013e3181e9322a. PMID 20664402
- [Background] Rolnik DL, O'Gorman N, Roberge S, Bujold E, Hyett J, Uzan S, Beaufils M, da Silva Costa F. Early screening and prevention of preterm pre-eclampsia with aspirin: time for clinical implementation. Ultrasound Obstet Gynecol. 2017 Nov;50(5):551-556. doi: 10.1002/uog.18899. No abstract available. PMID 28887883
- [Background] Shmueli A, Meiri H, Gonen R. Economic assessment of screening for pre-eclampsia. Prenat Diagn. 2012 Jan;32(1):29-38. doi: 10.1002/pd.2871. Epub 2012 Jan 11. PMID 22234821
- [Background] ACOG Committee Opinion No. 743 Summary: Low-Dose Aspirin Use During Pregnancy. Obstet Gynecol. 2018 Jul;132(1):254-256. doi: 10.1097/AOG.0000000000002709. PMID 29939936
- [Background] Tan MY, Wright D, Syngelaki A, Akolekar R, Cicero S, Janga D, Singh M, Greco E, Wright A, Maclagan K, Poon LC, Nicolaides KH. Comparison of diagnostic accuracy of early screening for pre-eclampsia by NICE guidelines and a method combining maternal factors and biomarkers: results of SPREE. Ultrasound Obstet Gynecol. 2018 Jun;51(6):743-750. doi: 10.1002/uog.19039. Epub 2018 Mar 14. PMID 29536574
- [Background] Akolekar R, Syngelaki A, Sarquis R, Zvanca M, Nicolaides KH. Prediction of early, intermediate and late pre-eclampsia from maternal factors, biophysical and biochemical markers at 11-13 weeks. Prenat Diagn. 2011 Jan;31(1):66-74. doi: 10.1002/pd.2660. PMID 21210481
- [Background] O'Gorman N, Wright D, Poon LC, Rolnik DL, Syngelaki A, Wright A, Akolekar R, Cicero S, Janga D, Jani J, Molina FS, de Paco Matallana C, Papantoniou N, Persico N, Plasencia W, Singh M, Nicolaides KH. Accuracy of competing-risks model in screening for pre-eclampsia by maternal factors and biomarkers at 11-13 weeks' gestation. Ultrasound Obstet Gynecol. 2017 Jun;49(6):751-755. doi: 10.1002/uog.17399. Epub 2017 May 14. PMID 28067011
- [Background] Crovetto F, Figueras F, Crispi F, Triunfo S, Pugia M, Lasalvia L, Chambers AE, Mills WE, Banerjee S, Mercade I, Casals E, Mira A, Rodriguez-Revenga Bodi L, Gratacos E. Forms of Circulating Luteinizing Hormone Human Chorionic Gonadotropin Receptor for the Prediction of Early and Late Preeclampsia in the First Trimester of Pregnancy. Fetal Diagn Ther. 2015;38(2):94-102. doi: 10.1159/000371516. Epub 2015 Feb 11. PMID 25676660
- [Background] Scazzocchio E, Figueras F, Crispi F, Meler E, Masoller N, Mula R, Gratacos E. Performance of a first-trimester screening of preeclampsia in a routine care low-risk setting. Am J Obstet Gynecol. 2013 Mar;208(3):203.e1-203.e10. doi: 10.1016/j.ajog.2012.12.016. Epub 2012 Dec 12. PMID 23246313
- [Background] Wright A, Wright D, Syngelaki A, Georgantis A, Nicolaides KH. Two-stage screening for preterm preeclampsia at 11-13 weeks' gestation. Am J Obstet Gynecol. 2019 Feb;220(2):197.e1-197.e11. doi: 10.1016/j.ajog.2018.10.092. Epub 2018 Nov 7. PMID 30414394
- [Background] Wright D, Gallo DM, Gil Pugliese S, Casanova C, Nicolaides KH. Contingent screening for preterm pre-eclampsia. Ultrasound Obstet Gynecol. 2016 May;47(5):554-9. doi: 10.1002/uog.15807. PMID 26643929
- [Background] Robinson HP, Fleming JE. A critical evaluation of sonar "crown-rump length" measurements. Br J Obstet Gynaecol. 1975 Sep;82(9):702-10. doi: 10.1111/j.1471-0528.1975.tb00710.x. PMID 1182090
- [Background] Figueras F, Meler E, Iraola A, Eixarch E, Coll O, Figueras J, Francis A, Gratacos E, Gardosi J. Customized birthweight standards for a Spanish population. Eur J Obstet Gynecol Reprod Biol. 2008 Jan;136(1):20-4. doi: 10.1016/j.ejogrb.2006.12.015. Epub 2007 Feb 6. PMID 17287065
- [Background] Committee Opinion No. 638: First-Trimester Risk Assessment for Early-Onset Preeclampsia. Obstet Gynecol. 2015 Sep;126(3):e25-e27. doi: 10.1097/AOG.0000000000001049. PMID 26287789
- [Derived] Trilla C, Luna C, De Leon Socorro S, Rodriguez L, Ruiz-Romero A, Mora Brugues J, Benitez Delgado T, Fabre M, Martin Martinez A, Ruiz-Martinez S, Llurba E, Oros D. First-Trimester Sequential Screening for Preeclampsia Using Angiogenic Factors: Study Protocol for a Prospective, Multicenter, Real Clinical Setting Study. Front Cardiovasc Med. 2022 Jul 26;9:931943. doi: 10.3389/fcvm.2022.931943. eCollection 2022. PMID 35958398

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT04767438/Prot_SAP_000.pdf